CLINICAL TRIAL: NCT03062397
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase IIa Clinical Trial to Evaluate the Efficacy and Safety of JPI-289 in Patients With Acute Ischemic Stroke
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of JPI-289 in Patients With Acute Ischemic Stroke
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JPI-289-P2
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — JPI-289

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low-dose group (Experimental): JPI-289 Low dose or placebo
  Interventions: Drug: JPI-289 Low-dose
- High-dose group (Experimental): JPI-289 High dose or placebo
  Interventions: Drug: JPI-289 High-dose
- Placebo group (Placebo Comparator): Same dosage of JPI-289 low and high dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JPI-289 Low-dose — JPI-289 Low dose will be intravenously administered during 24 hours
  Arms: Low-dose group
Drug: JPI-289 High-dose — JPI-289 High dose will be intravenously administered during 24 hours
  Arms: High-dose group
Drug: Placebo — Same dosage of JPI-289 Low and Hogh dose will be intravenously administered during 24 hours
  Arms: Placebo group

SUMMARY:
Clinical Trial to Evaluate the Efficacy and Safety of JPI-289 in Patients With Acute Ischemic Stroke

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute ischemic stroke, aging ≥ 19
* Confirmed to have acute anterior circulation cerebral artery occlusion in intracranial internal carotid artery (IICA) or middle cerebral artery (MCA) M1 segment by CT or MR angiography.
* National Institutes of Health Stroke Scale(NIHSS) is 6~30 before endovascular recanalization therapy (ERT)
* Subject who is reperfused with 2b or 3 stages of thrombolysis in cerebral infarction (TICI) (However, if angiography is conducted for thrombectomy after IV tPA treatment and the effect of tPA results in TICI 2b-3 reperfusion, the subject can participate)
* Subject who can administer IP within 6.5 hrs of symptom development
* Subject who can administer IP within 30 min of vascular reperfusion
* Subject who can evaluate MRI within 90 min of vascular reperfusion

Exclusion Criteria:

* Subject who is contraindicated for endovascular recanalization
* Subject who has hypersensitivity to contrast agent or component of investigational product
* Prohibited or unable to perform MRI test
* Medical history that is related to bleeding
* History of hemorrhagic stroke within 6 months of study participation
* Subjects with chronic liver disorder
* Kidney disorder (Serum creatinine > 3 mg/dL)
* Life expectancy is less than 3 months due to concomitant disease other than stroke
* Pregnant or lactating women
* Those who have taken tirofiban (anticoagulant agent) during endovascular recanalization therapy
* Those who have taken other investigational drugs and/or medical instruments 12 weeks prior to screening
* Subject is unable to be followed up
* Subject is deemed unable to participate the study in the opinion of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-12-09 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Infact growth ratio from baseline | 4 days from baseline

CONTACTS AND LOCATIONS:
Locations (15):
- South Korea (15):
  - Dong-A University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Yeungnam University Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Catholic Kwandong University International St. Mary'S Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Gyeongsang National University Hospital, Jinju
  - Pusan National University Hospital, Pusan
  - Ewha Womans University Seoul Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No